CLINICAL TRIAL: NCT07321314
Title: The Disease Burden of RSV Infection in Hong Kong
Brief Title: RSV Burden in Hong Kong
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ka Pang Chan, Professor, Chinese University of Hong Kong
Other Study IDs: RSV burden
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: RSV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Nasopharyngeal aspirate / swab, saliva, sputum, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RSV group: Patients with respiratory tract infection symptom and RSV confirmed in clinical specimens
  Interventions: Diagnostic Test: Serial specimen sampling
- Control group: Patients with respiratory tract infection symptom but no RSV confirmed in clinical specimens

INTERVENTIONS:
Diagnostic Test: Serial specimen sampling — Serial sampling of nasopharyngeal swab, saliva and sputum for RSV on day 3, 5, 7, 14, 28 (during hospitalization) for patients confirmed with RSV infection. Blood taking will be arranged on day 28 for serology purpose
  Groups: RSV group

SUMMARY:
RSV infection causes significant mortality and morbidity in susceptible adults. There are many publications on the global RSV disease burden in infants and young children but data on adults are lacking with lots of knowledge gaps. Currently there is no established effective antiviral therapy for RSV. RSV vaccines have recently become available commercially but the Center for Health Protection (Hong Kong) has yet to discuss procurement of RSV vaccines for the high risk groups. Thus a prospective study to assess the disease burden of RSV infection in adults would be of great interest.

DETAILED DESCRIPTION:
Respiratory syncytial virus (RSV) is an important cause of lower respiratory tract (LRT) infection in infants and young children, leading to hospitalizations and death. Its impact in adults has only been appreciated in recent years. Increasing evidence suggests that severe LRT RSV infections can occur, especially among the older adults and those with underlying comorbidities. RSV-related hospitalizations in adults, especially those older than 65 years, have increased markedly in the past decade. RSV was associated with longer hospitalization, more complications, higher mortality and hospitalization costs as great as influenza among older adults. RSV has accounted for 5-15% of community-acquired pneumonia, 10% of hospital admissions for acute cardiorespiratory diseases, and excessive deaths during seasonal peaks in adults. A systematic review in the UK has shown that RSV may have a substantial burden in UK adults. However, available data were limited and highly heterogenous, with further studies needed to characterise the burden of RSV in adults and to validate their findings. In a cross-sectional study over 5 RSV seasons in the US, 22% of hospitalized adults aged 50 years or older with RSV infection experienced an acute cardiac event (most frequently acute heart failure 16%), including 1 in 12 adults (8.5%) with no documented underlying cardiovascular disease. Acute cardiac events occurred more often among those with(33%) vs without(9%) underlying cardiovascular disease and were associated with nearly twice the risk of severe outcomes.

Over the last 2 decades, several retrospective and prospective studies based on nasopharyngeal (NP) swab PCR have examined the morbidity and mortality of RSV infection in HK. Among 4912 children hospitalized with RSV from 2009 to 2011, 118(2.4%) required paediatric ICU admission while chronic lung disease was the risk factor for the duration of PICU admission. Two retrospective studies showed that RSV mainly occurred in Spring and Summer in HK from April to September while RSV posed a heavy burden on children with heart disease. It was estimated the annual incidence of RSV infection requiring hospitalization as 2.5/1000 children <5 years old with a mortality of 0.15% among hospitalized cases. RSV conferred higher fatality than influenza and was the second killer among hospitalized elderly. In a retrospective study on 19,361 adult patients hospitalized for pneumonia, RSV infection was associated with higher mortality than influenza A or B (8.0% vs. 4.7% or 4.2%). The association with higher mortality in RSV persisted even in patients without chronic pulmonary disease or heart failure. Another retrospective cohort study was on all adults (≥18 years) with virologically confirmed RSV infection during 2009-2011 (N = 607) in comparisons to 547 adults hospitalized with seasonal influenza in the same period. RSV could cause severe LRT complications in older adults, resulting in respiratory failure, prolonged hospitalization, and high mortality similar to seasonal influenza while corticosteroids did not seem to improve outcomes. This retrospective study has shown that older age, radiographic evidence of pneumonia, need for ventilatory support, bacterial superinfection, elevated urea and elevated white cell count were independent risk factors associated with poorer survival.

The investigators published 3 prospective studies looking at the impact of RSV on acute exacerbations of chronic obstructive pulmonary disease (AECOPD), viral loads and cytokines/chemokines of adults with RSV infection. Among 505 admissions of AECOPD with nasopharyngeal aspirate (NPA) performed, 2.3% tested positive for RSV while paired serology showed 4-fold rise in viral titers in 2.2% of patients. A prospective study among adults hospitalized for PCR-confirmed RSV infections (n = 123) showed frequent occurrence of LRT complications causing respiratory failure (52.8%), requirement for assisted ventilation (16.3%), and ICU admission/death (12.2%). High viral RNA concentration was detected at time of hospitalization, including patients who presented within 2 days of illness (day 1-2, 7.29 ± 1.47; day 3-4, 7.28 ± 1.41; day 5-8, 6.66 ± 1.87 log10 copies/mL). RNA concentration was independently associated with risk of complications and respiratory failure (adjusted OR 1.40 per log10 copies/mL increase, 95%CI, 1.03-1.90; P = 0.034). Another prospective observational study in adults with RSV infection (71 hospitalized patients and 10 outpatients) showed that among the hospitalized adults, 61% required supplemental oxygen therapy, and 18% had severe disease requiring non-invasive ventilation (NIV) or intensive care, or died within 30 days. Inflammatory cytokine/chemokines IL-6, CXCL8/IL-8, CXCL9/MIG and CXCL10/IP-10 increased significantly during the acute phase of illness. IL-6 concentration was independently associated with severe disease after adjusting for confounding factors. In contrast to the study findings by Lee N et al, RSV viral load was not associated with disease severity throughout the clinical course in this prospective study of a smaller sample size.

While these retrospective and prospective studies based on NP swab PCR have provided some useful data on the morbidity and mortality of patients with confirmed RSV infection and in a specific COPD population, there is still lack of data from prospective studies on the disease burden of RSV in adults in HK. In addition, there is growing data that the sensitivity of PCR using NP swabs in diagnosing RSV is not as sensitive as using sputum or saliva PCR and serology. In a prospective cohort study over two study periods (2021 to 2022) of patients aged ≥ 40 years hospitalized for acute respiratory illness (ARI) in Louisville, KY., Ramirez J, et al found that among 1766 patients enrolled, 100% had NP swab, 99% saliva, 34% sputum, and 21% paired serology specimens. RSV was diagnosed in 56 (3.2%) patients by NP swab alone, and in 109 (6.2%) patients by NP swab plus additional specimens, corresponding to a 1.95 times higher rate [95% (CI) 1.62, 2.34]. Limiting the comparison to the 150 subjects with all four specimen types available (i.e., NP swab, saliva, sputum, and serology), there was a 2.60-fold increase (95% CI 1.31, 5.17) compared to NP swab alone (3.3% versus 8.7%). Sensitivities by specimen type were: NP swab 51%, saliva 70%, sputum 72%, and serology 79%. In a Korean study comparing the detection rates of respiratory viruses from NP swabs and sputum using a multiplex real-time reverse transcription-polymerase chain reaction (rtRT-PCR), adults who were admitted or presented to the clinics with acute respiratory symptoms were recruited from 1 Nov 2012 to 31 March 2013. The positive rate was 53% (81/154) for NP swabs and 68% (105/154) for sputum (P<0.001). Among 134 viruses identified for 107 illnesses, influenza A virus, RSV A, HRV, coronavirus OC43, and adenovirus were detected more frequently in sputum samples than in NP swabs (P<0.001). Importantly, 12 of 44 (27%) influenza A infections and 11 of 27 (41%) RSV infections were positive in only sputum samples.19 Wiseman DJ, et al. found that RSV infection was associated with 8.7% of AECOPD in their cohorts but confirmed that many infections would be missed with a reliance on PCR alone. RSV infection was identified as the cause of 27 of 310 attended exacerbations. Of these, were detected by PCR alone and 16 were detected exclusively by serology (an increase in RSV Nucleoprotein -specific antibody); 4 were detected by both methods. There was a higher positivity rate for RSV from sputum versus NP swabs (7.69% vs 2.02%, P=0.0061). Therefore, 59% of RSV associated AECOPD were negative on PCR despite a swab being obtained by highly trained staff within 5 days of symptom onset.

The investigators aim to study a) the incidence of RSV infection based on a statistical and economic model to estimate the annual incidence and healthcare cost of medically attended RSV disease among adults in HK; b) the risk factors associated with severe RSV infection.

The investigators hypothesize that the disease burden of RSV has been under-estimated by previous studies based on NP swab PCR and RSV causes significant morbidity and mortality in adults in addition to substantial healthcare expenses.

ELIGIBILITY:
Inclusion Criteria:

* Community-acquired respiratory tract infection symptoms
* Age >= 18

Exclusion Criteria:

* Unable to provide a good quality of sputum and saliva

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for community-acquired respiratory tract infection symptoms
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of RSV infection | 1 month
  The incidence of RSV infection based on the RSV detection rate in respiratory specimens collected from patients with respiratory tract infection symptoms

SECONDARY OUTCOMES:
Incidence of severe RSV infection | 1 month
  The incidence rate of severe RSV infection among patients with respiratory tract infection symptoms, as defined by NIV use, intensive care unit admission, or death

CONTACTS AND LOCATIONS:
Overall Officials: David SC Hui, MD, Study Director — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No